CLINICAL TRIAL: NCT02512770
Title: Esaphageal Balloon Dilatation in Children: Hemodynamic , Ventilatory Changes and Complications
Brief Title: Hemodynamic and Respiratory Effects of Esophageal Dilation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Ayse Cigdem Tutuncu (Other); Senol Emre (Unknown); Fatis Altindas (Unknown); Kaya, Guner, M.D. (Individual)
Responsible Party: Principal Investigator, pinar kendigelen, M.D.(Anesthesiology Specialist), Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 270718
Record Dates: First submitted 2015-07-26; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Obstruction of Esophagus; Respiratory Complication; Hemodynamic Instability
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dilatation (Experimental): esaphageal dilatation group
  Interventions: Procedure: endoscopic dilatation
- control (No Intervention): control group ( only endoscopy for control)

INTERVENTIONS:
Procedure: endoscopic dilatation
  Arms: dilatation

SUMMARY:
The aim of this study compares hemodynamic and respiratory changes and complications in children who undergoing endoscopy for esophageal balloon dilatation and endoscopy for only control.

DETAILED DESCRIPTION:
Esophageal strictures in children may develop as a secondary to a surgically repaired esophageal atresia (anastomatic strictures) or as a result of chemical injury after caustic ingestion. Emerging strictures are dilated with balloon catheter at regular intervals.

The possibility of various complications depending on the level of the stenosis during the dilation of esophagus. During Esophageal dilation may be pressed into airways and/or vascular structure.

ELIGIBILITY:
Inclusion Criteria:

* endoscopy for esaphageal dilatation and control
* ASA I-III
* 0-16 year old

Exclusion Criteria:

* ASA IV
* endoscopy for removing foreing body

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
peak inspiratory pressure | at time of endoscopy(0-40minute)

SECONDARY OUTCOMES:
complications ( laryngospasm, bronchospasm, can not be ventilated, decreased Sp02) | at time of endoscopy and after the endoscopy within 2 hours
Sp02 | at time of endoscopy and after the endoscopy within 2 hours
pressure levels for target tidal volume | at time of endoscopy(0-40minute)
mean arterial pressure-mmHg | at time of endoscopy(0-40minute)
heart rate-per/min | at time of endoscopy(0-40minute)

CONTACTS AND LOCATIONS:
Overall Officials: Guner Kaya, Prof., Study Director — Deapartment of Anesthesiology and Intensive Care, Cerrahpasa Medical Faculty,Istanbul University